CLINICAL TRIAL: NCT04173845
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Clinical Study of the Prevention of Levodopa-Induced Dyskinesia With Tianqi Pingchan Granule
Brief Title: Double Randomized and Placebo Controlled Trail of Tianqi Pingchan Granule to Prevent Levodopa-Induced Dyskinesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Affiliated Hospital of Nanjing University of Chinese Medicine (Other); Xin Hua Hospital of Zhejiang Province (Other); Suqian Branch, Jiangsu Province Hospital (Unknown); Huai'an First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XHEC-C-2019-033-2
Record Dates: First submitted 2019-11-05; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-10

CONDITIONS: Levodopa-Induced Dyskinesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tianqi Pingchan Granule group (Experimental): Tianqi Pingchan Granule were manufactured according to Good Manufacturing Practice (GMP) by Sichuan Neo-Green Pharmaceutical Technology Development Co., Ltd. , granule, twice a day, for six months.
  Interventions: Drug: Tianqi Pingchan Granule
- Tianqi Pingchan Granule Placebo group (Placebo Comparator): placebo, granule, twice a day, for six months.
  Interventions: Drug: Tianqi Pingchan Granule Placebo

INTERVENTIONS:
Drug: Tianqi Pingchan Granule — Tianqi Pingchan Granule are given twice a day
  Arms: Tianqi Pingchan Granule group
Drug: Tianqi Pingchan Granule Placebo — Tianqi Pingchan Granule Placebo
  Arms: Tianqi Pingchan Granule Placebo group

SUMMARY:
A randomized, double-blind, placebo-controlled multicenter clinical trial was used to observe the effectiveness, safety and side effects of Tianqi Pingzhan Granule in the prevention of levodopa induced dyskinesia, so as to determine the clinical efficacy of Tianqi Pingzhan Granule in the prevention of levodopa induced dyskinesia.

DETAILED DESCRIPTION:
The aim of this clinical trail is to evaluate the effect of Tianqi Pingzhan Granule in the prevention of levodopa induced dyskinesia in adults. All patients included in the study should meet the inclusion criteria. Half of participants will receive Tianqi Pingzhan Granule, while the other half will receive a placebo of Tianqi Pingzhan Granule. All participants will be assigned to either the active group or the control group randomly. During the clinical trail both doctors and patients are double-blind except serious adverse events occurred.

ELIGIBILITY:
Inclusion Criteria:

Patients with PD aged 30-85，have at least the following two conditions:

1. Dosage of Levodopa ≥ 400mg/d;
2. Grade of H&Y≥3;
3. risk score of dyskinesia>4;

Exclusion Criteria:

1. PD patients with dyskinesia;
2. Taking other Chinese medicines against Parkinson's disease;
3. pregnant and lactating women;
4. Impaired cognitive function (according to pre-entry MMSE score):

   secondary education level: MMSE <24 points; primary education level <20 points; illiterate <17 points;
5. accompanied by a history of mental illness;
6. impaired liver and kidney function;
7. accompanied by severe other systemic diseases;
8. Previous traditional Chinese medicine preparations or serious adverse reactions
9. Before the enrollment, the EKG showed obvious abnormalities and required clinical intervention.
10. PD related brain surgery
11. Patients who are participating in other clinical studies or has participated other clinical studies within 30 days before
12. Patients unable to cooperate with the survey

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
new dyskinesia attack | 48 weeks
  The occurrence of Levodopa-Induced dyskinesia

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 48 weeks
  Change in Unified Parkinson's Disease Rating Scale (MDS-UPDRS) total score of part III from Day 1 to 1 year. The part III of the MDS-UPDRS assess motor function in best on phase. The score range is 0-132, where a higher score means more severe motor impariment.
Patient diaries | 48 weeks
  Change in daily "OFF"-time as assessed with patient diaries from run-in to 48 weeks. This is a self administerd diary where patients assess their motor state every half hour during 24 hours.
MMSE（Mini-Mental State Examination） | 48 weeks
  To assess the degree of cognitive impairment of patients. The score range is 0-30, where a higher score means more severe cognitive impariment.
HAMA (Hamilton Anxiety Scale) | 48 weeks
  To assess the severity of anxiety symptoms. The score range is 0-56, where a higher score means more severe anxiety symptoms.
HAMD-24(Hamilton Depression Scale-24) | 48 weeks
  To assess the severity of depression symptoms. The score range is 0-96, where a higher score means more severe depression symptoms.
NMSQuest（Nonmotor symptoms Questionnaire） | 48 weeks
  To assess the severity and frequency of non-motor symptoms of Parkinson's disease. The score range of severity and frequency is 0-90 respectively, where a higher score means more severe and frequent non-motor symptoms of Parkinson's disease.
PDSS （Parkinson's Disease Sleep Scale） | 48 weeks
  To assess the severity of sleep of Parkinson's disease patients. The score range is 0-150, where a higher score means more severe sleep disorders.
ESS （Epwroth Sleepiness Scale） | 48 weeks
  To assess excessive daytime sleepiness in patients with Parkinson's disease. The score range is 0-24, where a higher score means more severe sleep disorders.
SCOP-AUT(scale for outcomes in Parkinson's disease for autonomic symptoms) | 48 weeks
  To assess the severity of autonomic symptoms. The score range is 0-104, where a higher score means more severe autonomic symptoms.
PD-ADL（Parkinson's disease-Activity of Daily Living Scale） | 48 weeks
  To assess the severity of Daily Living activity . The score range is 0-4, where a higher score means more severe daily living activity of Parkinson's disease patients.
Clinical Global Impression | 48 weeks
  Change score is an ordinal measure of change with a range of 0 (not assessed) to 7 (very much worse). A score of 4 is associated with "no change.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenguo Liu, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No